CLINICAL TRIAL: NCT05547061
Title: A Phase 1/2 Clinical Trial to Evaluate the Safety, Tolerability, Dosimetry, and Anti-tumor Activity of Ga-68-NGUL / Lu-177-DGUL in Patients With Metastatic Castration-resistant Prostate Cancer (mCRPC) Refractory to Standard Therapy
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Cellbion Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: Lu-PSMA001
Record Dates: First submitted 2022-09-13; First posted 2022-09-21 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Prostate Cancer; mCRPC
Keywords: PSMA
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Phase 1 Part A(Healthy/Disease group) (Experimental): Subjects are administered intravenously a single dose of 2MBq/kg of Ga-68-NGUL.
  Interventions: Drug: Ga-68-NGUL
- Phase 1 : Part B(Low dose) (Experimental): Subjects with positive lesions for Ga-68-NGUL are administered intravenously with low dose(150mCi) of Lu-177-DGUL.
  Interventions: Drug: Lu-177-DGUL; Drug: Ga-68-NGUL
- Phase 1 : Part B(High dose) (Experimental): Subjects with positive lesions for Ga-68-NGUL are administered intravenously with high dose(200mCi) of Lu-177-DGUL.
  Interventions: Drug: Lu-177-DGUL; Drug: Ga-68-NGUL
- Phase 2 (Experimental): Subjects with positive lesions for Ga-68-NGUL are administered intravenously with Lu-177-DGUL with the determined RP2D.
  Interventions: Drug: Lu-177-DGUL; Drug: Ga-68-NGUL

INTERVENTIONS:
Drug: Lu-177-DGUL — Administered intravenously once every 6 weeks (1 cycle) for a maximum of 6 cycles.
  Arms: Phase 1 : Part B(High dose); Phase 1 : Part B(Low dose); Phase 2
Drug: Ga-68-NGUL — Administered intravenously during screening and every 12 weeks after the first administration of Lu-177-DGUL.

SUMMARY:
This clinical trial is an open-label, single-arm, multi-center, escalation (Phase 1 Part B only), rater-blind (Phase 2 only), phase 1/2 trial to evaluate the diagnostic validity/safety of Ga-68-NGUL and efficacy/safety of Lu-177-DGUL on the anti-tumor activity that aims to simultaneously evaluate diagnostic and therapeutic validity.

ELIGIBILITY:
Inclusion Criteria:

* Male patients of 19 years or older
* Patients with metastatic diseases due to adenocarcinoma of the prostate as confirmed
* Patients whose blood testosterone levels at the screening visit meet the castration criteria(< 50 ng/dL)
* Patients with advanced metastatic castration-resistant prostate cancer who have failed standard treatment or no longer have standard treatment available
* Those who are maintaining androgen deprivation therapy (ADT) regardless of the type
* Patients receiving bone resorption treatment who have maintained a stable dose for at least 4 weeks prior to baseline
* Patients with positive lesions on Ga-68-NGUL PET scan
* Patients with Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
* Patients with an expected survival of 6months or more
* Patients with confirmed adequate hematological function, renal and hepatic function according to the following criteria
* Patients who have voluntarily consented to participate in this clinical trial and signed the informed consent form

Exclusion Criteria:

* Patients with hematologic malignancy, including lymphoma and solid cancers other than prostate cancer, within 3 years prior to baseline
* Patients who have received chemotherapy, biotherapy, or immunotherapy for prostate cancer treatment within 4 weeks prior to baseline
* Patients who have received radiation chemotherapy or radiation therapy within 12 weeks prior to baseline
* Patients who have received high-dose chemotherapy requiring hematopoietic stem cell therapy within 2 years prior to baseline
* Those who had previously received PSMA-targeted treatment or received radiopharmaceutical treatment, such as radium-223, within 6 months prior to baseline
* Patients with symptomatic central nervous system metastases
* Patients with unsuitable medical history or surgical/procedural history
* Patients with severe drug hypersensitivity and a history of hypersensitivity to the investigational product and similar drugs
* Patients receiving concomitant nephrotoxic drugs
* Patients with severe claustrophobia that is not controlled with anti-anxiety medications
* Patients with hypersensitivity reactions to components of the investigational product
* If the partner is a female of childbearing potential, patients who do not intend to abstain from abstinence or use appropriate contraceptive methods for at least 3 months after the end of the clinical trial period and investigational product administration
* Patients who have been administered with other investigational products or treated with clinical investigational devices within 4 weeks prior to baseline
* Patients who cannot participate in the clinical trial as determined by other investigators

Min Age: 19 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 91 (Actual)
Dates: Start 2021-04-12 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate(ORR) according to RECIST 1.1 | From baseline until radiographic progression or death from any cause, whichever comes first. assessed up to 36 months
  ORR is defined as the proportion of participants with best overall response of complete response or partial response according to RECIST 1.1

SECONDARY OUTCOMES:
PSA response rate(> 50% reduction compared to PSA before treatment) | baseline up to 24 weeks
  defined as the proportion of subjects who achieved a PSA response, which is considered a reduction of > 50% from baseline prior to treatment
PSA % change | baseline up to 24 weeks
  defined as the % change of PSA level compared to baseline.
PSA progression-free survival (PSA PFS) | From baseline until radiographic progression or death from any cause, whichever comes first. assessed up to 36 months
  from baseline until the time point at which PSA progression is confirmed or the time point of death is collected, whichever comes first.
Objective Response Rate(ORR) according to mPERCIST | baseline up to 24 weeks
  defined as the proportion of participants with best overall response of complete response or partial response according to RECIST 1.1
Best overall response(BOR) according to RECIST 1.1 and mPERCIST criteria | baseline up to 24 weeks
  defined as the best response among all responses at each time point from the start date of Lu-177-DGUL administration.
Waterfall plot according to best PSA response | baseline up to 24 weeks
  % change in PSA with the highest percentage decrease in PSA values from baseline.
Disease Control Rate(DCR) according to RECIST 1.1 and mPERCIST criteria | baseline up to 24 weeks
  defined as the proportion of participants with Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) according to RECIST v1.1.
Duration of Response(DOR) according to RECIST 1.1 and mPERCIST criteria | From baseline until radiographic progression or death from any cause, whichever comes first. assessed up to 36 months
  defined as the duration between the date of first documented Best Overall Response (BOR) of Complete Response (CR) or Partial Response (PR) and the date of first documented radiographic progression or death due to any cause.
PSA Doubling time | From baseline until radiographic progression or death from any cause, whichever comes first. assessed up to 36 months
  defined as the date of doubling time of PSA level from baseline.
Radiological progression-free survival (rPFS) | From baseline until radiographic progression or death from any cause, whichever comes first. assessed up to 36 months
  defined the date of first radiological evaluation of disease progression from the first day of administration of Lu-177-DGUL or the time of death, whichever comes first.
Waterfall plot according to tumor change rate | baseline up to 24 weeks
  The size of the target lesion (according to RECIST v1.1) and SUVpeak (according to mPERCIST) % change compared to the baseline are plotted as a waterfall plot
Overall survival (OS) | From baseline until radiographic progression or death from any cause, whicheve. assessed up to 36 months.
  defined as the date from the first day of administration of Lu-177-DGUL to death
Pain intensity (NRS) and opioid analgesic use | baseline up to 24 weeks
Quality of life (QOL): EORTC QLQ-C30, EORTC QLQ-PR25, EQ-5D-5L | baseline up to 24 weeks

CONTACTS AND LOCATIONS:
Locations (4):
- South Korea (4):
  - Chonnam National University Hwasun Hospital, Hwasun
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
  - Seoul National University Bundang Hospital, Seoul